# Study Protocol, NCT 03604497

(last updated 8/16/19)

## **Beacon Study Protocol**

#### I. Consent

There are two ways for participants to complete consent. Participants who scheduled an appointment are given the option to complete the consent and questionnaires before they come download the app. If they indicate they have done this method, **you must check on Qualtrics and make sure that they have completed this step before downloading the app on their phones.** If they have completed the consent and questionnaires, inform them about how the app functions and the purpose of the study and answer any questions they have.

Alternatively, we can complete consent in lab. Consent will be done using the iPads in lab if the participant is a walk-in appointment or if they did not complete consent before their appointment. Click on the "Beacon Consent" app on the iPads to continue. Enter the participant ID into the survey, which can be found on the "Beacon Participant List" Excel spreadsheet in the Shares Drive inside the "BEACON" Folder. Select the first available ID number.

Explain the consent form briefly to participants, allow them to read the consent for and answer any questions. Inform them about how the app functions and the purpose of the study. If they select "Agree", you may proceed.

#### II. Questionnaires

For participants who have not yet completed questionnaires, they should be completed in the waiting room on the iPads following completion of the consent process. Complete:

- Walking Journal
- Cell phone usage survey
- Demographics sheet

Collect iPads once participants have completed the survey.

### III. Download App

Participants who have finished the consent process and the surveys can bring their phones back for download. Ideally, while one researcher works with participants to download the app, another researcher can have participants fill out the W-9 form and process the payment.

## IV. Payment

Have participants complete W-9 form for payment. Greenphire will be used to process each participant's payment. Anyone with access to the Greenphire login can upload the participant's information to Greenphire. Log in from <a href="https://www.clincard.com/login/">https://www.clincard.com/login/</a>. Click on "Register Subject" and select the study ending with "300001917". Enter in participants' Subject ID, first and last name, address, and date of birth. Click on "Register". Click on "Assign Card". Click on "Request Payment".

Tell participants to allow about 24 hours for payment to be approved. Thank them for coming in and remind them of the following:

- 1. They should not delete the app off their phone for the full Fall semester. We will be monitoring this remotely and ask them to return to lab if they delete the app.
- 2. They should cross the intersection of 14<sup>th</sup> and University at least 4 times a week, and ideally more often.
- 3. If they have an iPhone and their phone goes dead (e.g. dead battery) or is turned off for some reason, they need to re-start the app. If they don't' do this, we will know it remotely and contact them to do it.
- 4. The app will not do anything for several weeks. At some point later in the semester, they will start getting alerts to remind them not to cross the street while distracted. We cannot tell them when these alerts will start, and it may be different for different people.